CLINICAL TRIAL: NCT03987672
Title: Study to Intervene With Nutrition for Gastroparesis
Acronym: SING
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment challenges
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Linda Nguyen, Clinical Associate Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 50803
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assess Nutritional Effects of Nutritional Formula (Other): Self-controlled study in which we will assess the nutritional effects of the Kate Farm Peptide 1.5 nutritional Formula in patients with gastroparesis, relative to their pre-enrollment nutritional formula regimen.
  Interventions: Dietary Supplement: Assess the nutritional effects of the Kate Farm Peptide 1.5 nutritional Formula

INTERVENTIONS:
Dietary Supplement: Assess the nutritional effects of the Kate Farm Peptide 1.5 nutritional Formula — Kate Farm Peptide 1.5 nutritional Formula
  Other Names: Study to Intervene with Nutrition for Gastroparesis

SUMMARY:
The study is a self-controlled study in which we will assess the nutritional effects of the Kate Farm Peptide 1.5 nutritional Formula in patients with gastroparesis, relative to their pre-enrollment nutritional diet regimen.

DETAILED DESCRIPTION:
The study is a prospective self-controlled study in which we will assess the nutritional effects of Kate Farm Peptide 1.5 nutritional formula in patients with gastroparesis, relative to their pre-enrollment diet regimen.

The duration of the study will be 12 weeks. We plan to recruit a total of 30 patients. Patients will undergo a baseline measurement of their height, weight, symptom burden, resting energy expenditure, inflammation, and microbiome. After study initiation, patient will undergo repeat testing at 1- and 3-months post-enrollment. Including the screening and baseline visits, there will be a total of 4 visits required to complete the study.

ELIGIBILITY:
Identify inclusion criteria.

* Male or female gender
* Ages 18 to 65
* Established diagnosis of gastroparesis confirmed by gastric emptying study within the last 5 years.
* No changes to gastroparesis medications in the 3 months prior to recruitment.
* Patients with hysterectomy, appendectomy, cholecystectomy and fundoplication are ok to participate.
* Able to give informed consent.
* Patient willing to supplement diet with Kate Farms
* Ability to adhere to the study visit schedule and other protocol requirements.

Identify exclusion criteria.

* Are nursing or pregnant.
* Diagnosis of mechanical small bowel obstruction within 3 months prior to recruitment
* Patients with a history of gastric surgery, including gastrectomy, small bowel resection or bariatric surgery
* The use of narcotic medications in the month prior to study enrollment or during the study period
* Diagnosis of short gut syndrome
* Allergic to any ingredients in the Kate Farms formula
* Untreated small intestinal bacterial overgrowth

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Gastroparesis Cardinal Symptom Index (GCSI) Symptoms Index (GCSI) score as measure of the effect of KF Peptide 1.5 nutritional formula. | Screening, Baseline and through end of study (12 weeks)
  9-item measure of severity of gastroparesis symptoms on a scale of 0-5 (none to worst)
  Higher values represent a worse outcome.

SECONDARY OUTCOMES:
Change in Patient Assessment of Gastrointestinal Disorders-Symptom Severity Index (PAGI-SYM) Disorders-Symptom Severity Index (PAGI-SYM) score as measure of the effect of KF Peptide 1.5 nutritional formula. | Baseline through end of study (12 weeks)
  20-item measure of upper gastrointestinal symptom severity on a scale of 0-5 (none to worst)
  Higher values represent a worse outcome.
Total energy requirement | At Baseline and end of study (12 weeks)
  Measurement of resting energy expenditure by indirect calorimetry
Inflammatory markers | Baseline through end of study (12 weeks)
  CRP C-reactive protein
Weight | Baseline through end of study (12 weeks)
  weight (kg)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Anh Nguyen, MD, Study Director — Stanford University
Locations (1):
- Stanford University School of Medicine, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No